CLINICAL TRIAL: NCT02830542
Title: A Phase 1b Randomized, Double-Blind, Placebo-Controlled, Ascending Single and Multiple Dose Study to Evaluate the Safety, Tolerability and Efficacy of SER-262 in Adults With Primary Clostridium Difficile Infection (CDI) to Prevent Recurrence
Brief Title: SER-262 Versus Placebo in Adults With Primary Clostridium Difficile Infection to Prevent Recurrence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Seres Therapeutics, Inc. (Industry)
Collaborators: Pharm-Olam International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SER-262-001
Record Dates: First submitted 2016-07-06; First posted 2016-07-13 (Estimated); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Clostridium Difficile Infection
Keywords: Clostridium difficile; C Diff; CDI
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SER-262 (Experimental): SER-262 [Single dose: 10(4), 10(5), 10(6), 10(7) or 10(8) SCFUs; Multiple dose 10(6), 10(7), or 10(8) SCFUs]
  Interventions: Drug: SER-262
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SER-262 — SER-262 is a rationally designed, multi-strain Ecobiotic® microbiome therapeutic produced synthetically by in vitro fermentation. It is a consortium of anaerobic, commensal bacteria in spore form, encapsulated for oral administration.
  Other Names: Cultivated Eubacterial Spore Suspension, Encapsulated
  Arms: SER-262
Drug: Placebo — Placebo will be identical to the investigational product but will not contain product spores or non-spore solids. Placebo will consist of 92% glycerol and 8% normal saline.
  Arms: Placebo

SUMMARY:
The study will involve administering a single dose of investigational drug or placebo in ascending dose cohorts. This study is designed to evaluate the safety and tolerability of investigational drug as well as the efficacy of investigational drug versus placebo in adults with primary (first episode) Clostridium difficile infection (CDI).

DETAILED DESCRIPTION:
SER-262-001 is a Phase 1b, randomized, double blind, placebo-controlled, ascending single dose clinical study with 2 treatment arms (SER-262 or placebo) in up to 8 dose cohorts. Patients who have been diagnosed with their first (primary) episode of CDI, defined as diarrhea (≥ 3 unformed stools per day for 2 consecutive days), a positive C. difficile stool test and who have responded to standard-of-care antibiotic will receive investigational drug or placebo on Day 1.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, indicating that the subject understands the purpose of and procedures required for the study.
2. Male or female subjects ≥ 18 years.
3. A primary (first) episode of CDI with documentation of the episode including CDI date, test results, antibiotic treatment (including start and stop dates), and response to treatment

Exclusion Criteria:

1. Females who are pregnant, breastfeeding, lactating, or planning to become pregnant during the study.
2. Known or suspected toxic megacolon and/or known small bowel ileus.
3. Active irritable bowel syndrome with diarrhea within the previous 12 months.
4. Major gastrointestinal surgery (eg, significant bowel resection or diversion) within 3 months before enrollment (this does not include appendectomy or cholecystectomy) or any history of total colectomy or bariatric surgery.
5. History of inflammatory bowel disease (ulcerative colitis, Crohn's disease, microscopic colitis) with diarrhea believed to be caused by active inflammatory bowel disease in the past 12 months.
6. Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73m2
7. Admitted to or expected to be admitted to an intensive care unit for medical reasons (not just boarding). Patients discharged from an intensive care unit before Day 1 may be enrolled.
8. Concurrent intensive induction chemotherapy, radiotherapy, or biologic treatment for active malignancy (patients on maintenance chemotherapy may only be enrolled after consultation with medical monitor).
9. Absolute neutrophil count < 500 cells/mm3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of SER-262 as assessed by incidence of AEs, lab results, vital signs, ECG, and physical examination findings | Up to 24 weeks after treatment
Relative risk of recurrence based on the proportion of subjects experiencing CDI recurrence in each SER-262 cohort compared to placebo up to 8 weeks after treatment | Up to 8 weeks after treatment

SECONDARY OUTCOMES:
Time to recurrence of CDI | Up to 24 weeks after treatment
Relative risk of recurrence of CDI up to 4, 12, and 24 weeks after treatment | Up to 4, 12, and 24 weeks after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michele Trucksis, PhD, MD, Study Director — Seres Therapeutics
Locations (22):
- United States (22):
  - North Alabama Research Center, LLC, Athens, Alabama
  - Lalla-Reddy Medical Corporation, Fountain Valley, California
  - eStudySite, La Mesa, California
  - San Marcus Research Clinic, Inc., Miami, Florida
  - Omega Research Consultants, Orlando, Florida
  - Emory University Hospital, Atlanta, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Snake River Research, Idaho Falls, Idaho
  - Anne Arundel Health System Research Institute, Annapolis, Maryland
  - Henry Ford Health System, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Sundance Clinical Research, LLC, St Louis, Missouri
  - Mercury St. Medical Group, Butte, Montana
  - Quality Clinical Research, Omaha, Nebraska
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - University of Rochester Medical Center, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - Remington Davis, Columbus, Ohio
  - Regional Infectious Diseases & Infusion Center, Lima, Ohio
  - Baylor Scott & White Research Institute, Temple, Texas
  - Dr. Hansen Internal Medicine, Bountiful, Utah
  - Infectious Disease Associates of Central Virginia, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: No